CLINICAL TRIAL: NCT06270836
Title: A Prospective, Randomized, Double-masked, Sham-controlled, Multi-center, Two-arm, Phase 3 Study to Evaluate the Efficacy and Safety of Intravitreal Tarcocimab Tedromer in Participants With Diabetic Retinopathy (DR) - GLOW2
Brief Title: A Study to Evaluate the Efficacy and Safety of Tarcocimab Tedromer Compared With Sham Treatment in Participants With Diabetic Retinopathy (DR)
Acronym: GLOW2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kodiak Sciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KS301P108
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic Retinopathy; NPDR; KSI-301; VEGF; Anti-VEGF; Vascular Endothelial Growth Factor; Antibody Biopolymer Conjugate; Retinal Degeneration; Retinal Diseases; Eye Diseases; Retinopathy; Vision Disorders; Kodiak; Tarcocimab Tedromer; Tarcocimab; Diabetic Eye Disease
MeSH Terms: conditions — Diabetic Retinopathy; Retinal Degeneration; Retinal Diseases; Eye Diseases; Vision Disorders | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 into one of two arms: KSI-301 or sham.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: To preserve masking, 2 investigators are required for this study. The masked investigator will be responsible for examinations and safety assessments. The unmasked investigator will perform the injections and post-treatment assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tarcocimab 5 mg (Treatment Group A) (Experimental): Tarcocimab 5 mg via intravitreal injection at Day 1, Week 4, Week 8, Week 20, and Week 44.
  Interventions: Drug: Tarcocimab
- Treatment Group B (Sham Comparator): Sham injection on the same schedule as Treatment Group A
  Interventions: Other: Sham injection

INTERVENTIONS:
Drug: Tarcocimab — Intravitreal injection
  Other Names: Tarcocimab tedromer; KSI-301
  Arms: Tarcocimab 5 mg (Treatment Group A)
Other: Sham injection — The sham injection is a procedure that mimics an intravitreal injection. It involves pressing the blunt end of an empty syringe (without a needle) against the anesthetized eye. It is performed to maintain masking of the study.
  Arms: Treatment Group B

SUMMARY:
This study will demonstrate that tarcocimab 5 mg is superior to sham treatment in participants with DR.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-masked, two-arm, multi-center Phase 3 study to demonstrate that tarcocimab 5 mg is superior to sham treatment, with respect to the proportion of eyes improving from baseline at Week 48 in participants with DR.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to participation in the study.
* Type 1 or 2 diabetes mellitus and HbA1c of ≤12%.
* DR in the Study Eye (DRSS as determined by the reading center based on color fundus photographs), who have not previously received intravitreal medications for DR or DME, and in whom pan-retinal photocoagulation (PRP) can be safely deferred for at least 6 months per the Investigator.
* CST ≤320 microns and a BCVA ETDRS letter score in the Study Eye of ≥69 letters (approximate Snellen equivalent of 20/40 or better) in the Study Eye at screening and confirmed at Day 1; OR
* CST >320 and ≤350 microns and a BCVA ETDRS letter score in the Study Eye of ≥79 letters (approximate Snellen equivalent of 20/25 or better) in the Study Eye at screening and confirmed at Day 1.

Exclusion Criteria:

* Prior PRP in the Study Eye.
* Current anterior segment neovascularization (ASNV), vitreous hemorrhage, or tractional retinal detachment in the Study Eye.
* Prior intravitreal anti-VEGF treatment in the Study Eye for DR or DME within the last twelve (12) months prior to Day 1.
* Prior intravitreal or periocular steroid in the Study Eye for DR or DME within the last twelve (12) months prior to Day 1.
* Prior use of an investigational intravitreal treatment for DR or DME in the Study Eye.
* History of vitreoretinal surgery in the Study Eye.
* History of uveitis in either eye.
* Cataract in the Study Eye that in the judgment of the Investigator is expected to require surgical extraction within 12 months of screening.
* Significant media opacities, including cataract, in the Study Eye that might interfere with visual acuity, assessment of safety, OCT, or FP.
* Any history or evidence of a concurrent ocular condition present in the Study Eye, that in the opinion of the Investigator could require either medical or surgical intervention or alter visual acuity during the study.
* Active or suspected ocular or periocular infection or inflammation.
* Women who are pregnant or lactating or intending to become pregnant during the study.
* History of a medical condition that, in the judgment of the Investigator, would preclude scheduled study visits, completion of the study, or a safe administration of investigational product.
* Recent history (within the 6 months prior to screening) of myocardial infarction, stroke, transient ischemic attack, acute congestive heart failure or any acute coronary event.
* Uncontrolled blood pressure defined as a systolic value ≥ 180 mmHg or diastolic value ≥ 100 mmHg while at rest.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of eyes improving ≥2 steps on the Early Treatment Diabetic Retinopathy Diabetic Retinopathy Severity Scale (ETDRS DRSS) | Day 1 to Week 48
  Early Treatment Diabetic Retinopathy Diabetic Retinopathy Severity Scale (ETDRS DRSS), on a scale from 10 to 90, where lower scores represent better outcomes.

SECONDARY OUTCOMES:
Proportion of eyes developing a Sight-Threatening Complication(s) of diabetic retinopathy | Day 1 to Week 48
  Sight-threatening complications include diabetic macular edema, new or worsening proliferative diabetic retinopathy, and anterior segment neovascularization
Proportion of eyes improving ≥3 steps on Early Treatment Diabetic Retinopathy Diabetic Retinopathy Severity Scale (ETDRS DRSS) | Day 1 to Week 48
  Early Treatment Diabetic Retinopathy Diabetic Retinopathy Severity Scale (ETDRS DRSS), on a scale from 10 to 90, where lower scores represent better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Velazquez-Martin, MD, Study Director — Kodiak Sciences Inc
Locations (38):
- United States (37):
  - Retina Associates SW, Tucson, Arizona
  - Retina Consultants of Orange County, Fullerton, California
  - Global Research Management, Inc. - Lugene Eye Institute, Glendale, California
  - Retinal Consultants Medical Group, Inc., Modesto, California
  - Retina Consultants of Southern California, Redlands, California
  - Retinal Consultants Medical Group, Inc., Sacramento, California
  - Retina Group of New England, PC, Waterford, Connecticut
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Springfield Clinic LLP, Springfield, Illinois
  - Associated Vitreoretinal and Uveitis Consultants, Carmel, Indiana
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Retina Consultants of Nevada, Henderson, Nevada
  - Envision Ocular, LLC, Bloomfield, New Jersey
  - Asheville Eye Associates, Asheville, North Carolina
  - North Carolina Retina Associates (Cary), Cary, North Carolina
  - North Carolina Retina Associates (Wake Forest), Wake Forest, North Carolina
  - Cascade Medical Research Institute, Springfield, Oregon
  - Erie Retina Research, Erie, Pennsylvania
  - Charleston Neuroscience Institute, Charleston, South Carolina
  - Charles Retina Institute, Germantown, Tennessee
  - Southeastern Retina Associates PC, Knoxville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Panhandle Eye Group, LLP. - Southwest Retina Specialists, Amarillo, Texas
  - Austin Retina Associates, PLLC (Austin), Austin, Texas
  - Austin Research Center for Retina, Austin, Texas
  - Retina Consultants of Texas (Bellaire), Bellaire, Texas
  - Star Vision Research, Burleson, Texas
  - Retina Consultants of Texas (Katy), Katy, Texas
  - Texas Retina Associates, Plano, Texas
  - Austin Retina Associates, PLLC (Round Rock), Round Rock, Texas
  - Retina Consultants of Texas (San Antonio), San Antonio, Texas
  - Retina Consultants of Texas (Woodlands), The Woodlands, Texas
  - Piedmont Eye Center, Lynchburg, Virginia
  - Pacific Northwest Retina (Bellevue), Bellevue, Washington
  - Spokane Eye Clinical Research, Spokane, Washington
- Emanuelli Research & Development Center, LLC, Arecibo, Puerto Rico